CLINICAL TRIAL: NCT05601986
Title: Investigation of the Effect of Motor Imagery on Gait and Balance Functions in Children With Duchenne Muscular Dystrophy
Brief Title: Motor Imagery on Children With DMD on Gait and Balance Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gülsena Utku (Other)
Responsible Party: Sponsor-Investigator, Gülsena Utku, Principal Investigator, Halic University
Organization: Halic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MI on DMD
Record Dates: First submitted 2022-10-20; First posted 2022-11-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Gait; Balance; Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Physical Therapy Modalities; Rehabilitation; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy and Rehabilitation Program (Other): Control Group
  Interventions: Other: Physiotherapy and Rehabilitation Program
- Additional Motor Imagery Training to Physiotherapy and Rehabilitation Program (Experimental): Intervention Group
  Interventions: Other: Physiotherapy and Rehabilitation Program; Other: Additional Motor Imagery Training to Physiotherapy and Rehabilitation Program

INTERVENTIONS:
Other: Physiotherapy and Rehabilitation Program — The program will be held for 8 weeks, 2 days a week, with 40-minute sessions. Relaxation phase: Progressive relaxation. Stretching phase: Stretching exercises for the muscles of the gastrocnemius, hamstrings, hip flexors, hip adductors Strengthening phase: Isometric strengthening exercises for the tibialis anterior, quadriceps, hip extensors, and hip abductors muscles.
  Balance training phase: Two legs, one leg, balance with eyes open and eyes closed.
  Weight-bearing phase: Weight transfer to the front, back, and sides using the balance board.
  Other Names: Control group
Other: Additional Motor Imagery Training to Physiotherapy and Rehabilitation Program — The program will be held for 8 weeks, 2 days a week, with 40-minute sessions. Relaxation phase, Stretching phase, Strengthening phase,Balance training phase and Weight-bearing phase. Additional to the Physiotherapy and Rehabilitation Program, the Additional Motor Imagery Training program will be carried out for 8 weeks, 2 days a week, in addition to the 40-minute physiotherapy and rehabilitation program, accompanied by 25-30 minutes of supervision. It will be conducted by the researcher on two non-consecutive days of the week, by making appropriate appointments for the participants. During the program, participants will be asked to be in a quiet room. Sessions will consist of 4 consecutive phases: video watching, relaxation, motor imagery, and return to the environment.
  Other Names: Intervention group
  Arms: Additional Motor Imagery Training to Physiotherapy and Rehabilitation Program

SUMMARY:
The most common muscular dystrophy among pediatric neuromuscular diseases is Duchenne Muscular Dystrophy (DMD). There is no consensus on a standardized physiotherapy and rehabilitation program or exercise prescription in DMD. Motor imagery (MI) is defined as visualizing motor activities in one's mind without performing any movement. There are studies examining the effectiveness of motor imagery in stroke, cerebral palsy, Parkinson's, peripheral facial paralysis, and phantom pain. This study is aimed to examine the effect of motor imagery on gait and balance functions in children with Duchenne Muscular Dystrophy. Boys residing in Istanbul Turkey, between the ages of 5 and 12, with a diagnosis of DMD who have not lost their ability to ambulate independently will be included in the study. The included individuals will be divided into two groups due to randomization: Group A (Control Group Physiotherapy and Rehabilitation Program) and Group B (Additional Motor Imagery Training to Intervention Group Physiotherapy and Rehabilitation Program). While the physiotherapy and rehabilitation program is applied to the participants in Group A with 40-minute sessions on 2 non-consecutive days of the week for 8 weeks, the participants in Group B will receive an additional 25-30-minute motor imagery program to the physiotherapy and rehabilitation program. Participants were tested with Kinovea Gait Analysis, Timed Up and Go Test, 2 Minute Walking Test, Motor Function Rating Scale for Neuromuscular Diseases, timed performance tests, Pediatric Berg Balance Scale, Pediatric Fear of Fall Questionnaire (Ped-FOF) before and after the program. will be evaluated later. IBM SPSS (Statistical Package for Social Sciences) statistical program version 22.0 will be used for statistical analysis. The conformity of the variables to the normal distribution will be determined by the "Shapiro-Wilk Test". If the variables show normal distribution, the variation within the group will be analyzed with the "Paired Sample T Test", if not, the "Wilcoxon Test" will be analyzed. In the comparison between groups, if the variables show normal distribution, it will be done with the "Independent T Test" in independent groups and the "Mann Whitney U Test" if they do not show normal distribution. Categorical data distributions will be evaluated with the "Chi-square test". In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician-prescribed diagnosis of Duchenne Muscular Dystrophy
* Not having any injury or surgical operation in the last 6 months
* Being between Levels 1-5 (children who continue to ambulate independently) according to - Brooke Lower Extremity Functional Classification Modified Mini-Mental Test score >27
* Having the level of cooperation to follow the physiotherapist's instructions
* Volunteering to participate in research

Exclusion Criteria:

* Having severe contractures that interfere with functional activities
* Level 6-10 (children not capable of independent ambulation) according to the Brooke Lower Extremity Functional Classification
* To receive applications in addition to the physiotherapy and rehabilitation program or different from the physiotherapy and rehabilitation program

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
gait analysis1 | one week before the intervention and one week after the intervention
  Change from Baseline Stride length in meters
gait analysis2 | one week before the intervention and one week after the intervention
  Change from Baseline stride width in meters
gait analysis3 | one week before the intervention and one week after the intervention
  Change from Baseline Systolic cadence
gait analysis4 | one week before the intervention and one week after the intervention
  Change from Baseline walking speed in meters/second
balance | one week before the intervention and one week after the intervention
  Change from Baseline Pediatric Balance Scale in grades 0-56 points

SECONDARY OUTCOMES:
muscle strength measurement | one week before the intervention and one week after the intervention
  Strength measurements of lower extremity muscles

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Razak Özdinçler, Prof, Study Director — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No